CLINICAL TRIAL: NCT01424436
Title: Modulation of Beta-amyloid Levels in CSF and Plasma by GSK933776 in Patients With Mild Alzheimer's Disease or Mild Cognitive Impairment
Brief Title: Modulation of Abeta Levels by GSK933776 in Alzheimer's Disease Patient
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 113043
Record Dates: First submitted 2011-08-04; First posted 2011-08-29 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Alzheimer's Disease
Keywords: CSF sampling; Alzheimer's disease; Amyloid beta levels
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- GSK933776 1mg/kg (Experimental): single dose
  Interventions: Biological: GSK933776
- GSK933776 0.1 or 3mg/kg (Experimental): single dose
  Interventions: Biological: GSK933776
- GSK933776 3 or 6mg/kg (Experimental): single dose
  Interventions: Biological: GSK933776

INTERVENTIONS:
Biological: GSK933776 — 1mg/kg dose group
  Arms: GSK933776 1mg/kg
Biological: GSK933776 — 3mg/kg dose group
  Arms: GSK933776 0.1 or 3mg/kg
Biological: GSK933776 — 6mg/kg dose group
  Arms: GSK933776 3 or 6mg/kg

SUMMARY:
Modulation of beta-amyloid levels in CSF and plasma by GSK933776 in patients with mild Alzheimer's disease or mild cognitive impairment

DETAILED DESCRIPTION:
This is a phase I, an open label, single dose and parallel group study to assess short term pharmacodynamics and safety of GSK933776. The effect on the beta amyloid levels will be assessed in early (MCI) and mild Alzheimer's disease (AD) patients after a single dose of GSK933776 by i.v. administration.

ELIGIBILITY:
Inclusion Criteria:

* Probable mild Alzheimer's disease (MMSE 20-26) or mild cognitive impairment
* Increase in total tau or p-tau in CSF
* Decrease in amyloid beta in CSF
* Stable dose of cholinesterase inhibitors, memantine or selegine or no treatment
* Body weight less than 120 kg
* Willingness to comply with contraceptive methods if self or partner is of child-bearing potential

Exclusion Criteria:

* Any other cause of dementia
* Other significant neurologic or psychiatric illness
* Hachinski Ischemia Score >4
* More than 3 microbleeds on MRI
* Type 2 diabetes not controlled by diet
* Risk of cerebrovascular disease, cerebral haemorrhage or stroke
* History of systemic autoimmune disease
* Use of platelet anti-aggregates or anti-coagulants (Aspirin up to 325 mg/day is allowable)
* Use of chronic corticosteroids
* Uncontrolled hypertension in spite of antihypertensive medications
* Renal or hepatic insufficiency or clinically significant anaemia
* In nursing home care
* Contraindications to lumbar puncture or MRI
* Prior participation in therapeutic studies only after adequate wash-out period

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2011-12-08 (Actual); Study Completion 2011-12-08 (Actual)

PRIMARY OUTCOMES:
The temporal changes of amyloid beta levels in CSF after GSK933776 single dose administration in the patients with Alzheimer's disease and Mild Cognitive impairment | 22 hours
  To compare the changes of amyloid beta levels between the baseline (9 hours) and after single dose of GSK933776 iv administration of 13 hours

SECONDARY OUTCOMES:
The temporal changes of total and free amyloid beta levels in plasma after GSK933776 single dose administration in the patients with Alzheimer's disease and Mild Cognitive impairment | Two months
The temporal changes of Tau and phosphor Tau - 181 levels in CSF after GSK933776 single dose administration in the patients with Alzheimer's disease and Mild Cognitive impairment | 22 hours
Estimated pharmacokinetic parameters of AUC, Cmax and Tmax in CSF and plasma at multiple time points with various intervals. | three months
To assess the safety and tolerability after single dose of GSK933776 administration. | three months
  The safety and tolerability measures are performed at screening, dosing day and follow up. The assessments included: • Adverse event reporting and safety laboratory data. • CNS Safety: MRI and MMSE. • CVS safety: ECG and vital signs. •Anti-GSK933776 antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Germany (5):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
- Sweden (2):
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Andreasen N, Simeoni M, Ostlund H, Lisjo PI, Fladby T, Loercher AE, Byrne GJ, Murray F, Scott-Stevens PT, Wallin A, Zhang YY, Bronge LH, Zetterberg H, Nordberg AK, Yeo AJ, Khan SA, Hilpert J, Mistry PC. First administration of the Fc-attenuated anti-beta amyloid antibody GSK933776 to patients with mild Alzheimer's disease: a randomized, placebo-controlled study. PLoS One. 2015 Mar 19;10(3):e0098153. doi: 10.1371/journal.pone.0098153. eCollection 2015. PMID 25789616
- [Derived] Leyhe T, Andreasen N, Simeoni M, Reich A, von Arnim CA, Tong X, Yeo A, Khan S, Loercher A, Chalker M, Hottenstein C, Zetterberg H, Hilpert J, Mistry P. Modulation of beta-amyloid by a single dose of GSK933776 in patients with mild Alzheimer's disease: a phase I study. Alzheimers Res Ther. 2014 Apr 9;6(2):19. doi: 10.1186/alzrt249. eCollection 2014. PMID 24716469
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113043 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113043?search=study&search_terms=113043#rs
- Available data/document: Study Protocol: 113043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113043 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register